CLINICAL TRIAL: NCT05338697
Title: Validation of Early Prognostic Data for Recovery Outcome After Stroke for Future, Higher Yield Trials
Acronym: VERIFY
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: University of California, Los Angeles (Other); University of Auckland, New Zealand (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Pooja Khatri, Professor & Chair of Neurology, Yale University
Other Study IDs: G200291
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic
Keywords: VERIFY
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Ischemic & Hemorrhagic stroke patients: up to 657 stroke patients
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Diagnostic Test: Transcranial Magnetic Stimulation (TMS) — No intervention used. This study is using TMS to obtain motor evoked potential (MEP), a prognostic biomarker. The TMS procedure is being conducted during the first week of hospitalization, which required registration under an IDE. Only TMS devices that have received 510(k) clearance from the FDA are used in this study, consisting of MEGA-TMS and MagStim 200-2.

SUMMARY:
VERIFY will validate biomarkers of upper extremity (UE) motor outcome in the acute ischemic stroke window for immediate use in clinical trials, and explore these biomarkers in acute intracerebral hemorrhage. VERIFY will create the first multicenter, large-scale, prospective dataset of clinical, transmagnetic stimulation (TMS), and MRI measures in the acute stroke time window.

DETAILED DESCRIPTION:
Currently, 7 million US stroke survivors have significant disability, more than half with residual motor deficits. Motor function, particularly of the upper extremity (UE), is critical for regaining independence after stroke. UE function largely depends on integrity of motor cortex and its descending fibers, collectively termed the corticomotor system (CMS). Validated, clinically relevant biomarkers that identify biologically distinct patient subgroups are critically needed, particularly for the often affected and functionally important CMS. Their absence is a major obstacle to developing and personalizing new recovery therapies, especially in the early days post stroke.

Presence or absence of motor evoked potential (MEP) responses to TMS and extent of MRI-measured acute lesion load involving corticospinal tract (CST) are ready for formal validation. Also, the Predict Recovery Potential (PREP)-2 prediction tool, which sequentially combines acute clinical information and MEP status, is primed for multi-site validation.

The central objective is to validate the most biologically relevant and primed biomarkers of 90-day UE motor outcomes after ischemic stroke in the first large-scale, prospective, acute dataset of clinical, TMS, and MRI measures. The central hypothesis is that patients have different UE outcomes depending on CMS function measured with TMS, and on CST injury measured with MRI.

The specific aims are:

1. to externally validate the relationships that TMS and MRI biomarkers of CMS integrity have with 90-day UE motor impairment outcome and
2. to externally validate the PREP2 prediction tool to predict 90- day UE functional outcome. The study will also explore these biomarkers in acute intracerebral hemorrhage.

The study will comprehensively measure UE outcomes 90 days post-stroke in three domains of motor performance -impairment, function, and use - identified by the World Health Organization International Classification of Functioning, Disability and Health.

By establishing biomarkers for use in the acute stroke period to identify patient subgroups with distinct 90-day outcomes, the study will improve the efficiency of stroke recovery trials and inform rehabilitation decision-making.

Sample Size: up to 657 participants with complete biomarker data enrolled at up to 45 sites.

Trial Status: VERIFY received formal FDA IDE approval in November 2020 and received NIH funding in September 2021. Participating sites from the United States have been identified, and the study is now enrolling eligible participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Unilateral symptomatic stroke due to ischemia. (Note: Bilateral acute stroke is permitted if the stroke that is contralateral to the index stroke is asymptomatic).
3. Motor deficits in the acutely affected UE, defined as a Shoulder Abduction and Finger Extension (SAFE) score ≤ 8 out of 10 points20,61 (i.e., excluding full or nearly full motor strength in both shoulder abduction and finger extension) within 48 to 96 hours of stroke onset (or time last known well).

   a. Please note that, if significant imbalance is observed in SAFE score or MEP+ rates, the enrollment threshold for SAFE score may be updated with a formal study memo.
4. Provision of signed and dated informed consent form within 24 to 96 hours of stroke onset, (or time last known well). Note: Participant is considered "enrolled" upon starting TMS (at least one stimulation is delivered) or starting study-specific MRI pulse sequence (at least one MRI beep occurs)
5. Stated willingness to comply with all study procedures and availability for the duration of the study, including Day 90 visit which must occur in-person.
6. Fluent in study approved languages (i.e., English or Spanish)

Exclusion Criteria:

1. UE injury or conditions on paretic side that limited use prior to the stroke
2. Legally blind
3. Dense sensory loss on paretic side indicated by a score of 2 on NIHSS sensory item
4. Unable to abduct the shoulder or extend the fingers of the non-paretic UE on verbal command
5. Isolated cerebellar stroke
6. Symptomatic stroke in any location within 30 days prior to index stroke.
7. Co-enrollment in a trial of an intervention targeting the incident stroke (acute treatment or rehabilitation/recovery intervention) after baseline assessments for VERIFY are initiated
8. Known or expected inability to maintain follow-up with study procedures through 90 days
9. Cognitive or communication impairment precluding informed consent by the participant.
10. Major medical, neurological, or psychiatric condition that would substantially affect functional status
11. Non-cerebrovascular diagnosis associated with unlikely survival at 90 days
12. Pregnancy
13. Contraindication to noncontrast MRI (certain metallic implants, metallic foreign bodies or severe claustrophobia)
14. Contraindication to TMS

    1. Implanted electronic cardiac devices (e.g., Automatic Implantable Cardioverter-Defibrillator [AICD] or pacemaker)
    2. Any electronic devices in the body at or above the level of the seventh cervical vertebra (such as cochlear implant, cortical stimulator, deep brain stimulator, vagus nerve stimulator, cervical spine epidural stimulator, or ventriculoperitoneal shunt)
    3. Ferromagnetic intracranial metallic implant
    4. Skull defect related to current stroke
    5. Seizure after onset of current stroke
    6. Seizure within the last 12 months while taking anti-epileptic medications
    7. Previous serious adverse reaction to TMS
15. Anticipated inability to perform study procedures within 168 hours of symptom onset

    1. Unable to perform behavioral assessments within 48-120 hours of symptom onset (or time last known well).
    2. Unable to receive TMS within 72-168 hours or get MRI within 48-168 hours of symptom onset (or time last known well).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke consented within 24-96 hours of stroke onset in the acute hospitalization setting
Sampling Method: Non-Probability Sample
Enrollment: 657 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity-Fugl Meyer (UE-FM) for AIM 1 | 90 days post-stroke
  UE-FM score, as a continuous scale, adjusted for baseline score in analysis
Action Research Arm Test (ARAT) for AIM 2 | 90 days post-stroke
  ARAT categorized as 'excellent', 'good', 'limited', or 'poor'

OTHER OUTCOMES:
Motor Activity Log (MAL) | 90 days post-stroke
  MAL categorized as 0 to 3 versus >/=3 to 5.
modified Rankin Score (mRS) | 90 days post-stroke
  mRS level (0-6)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khatri, MD, Principal Investigator — Yale University; Steve Cramer, MD, Principal Investigator — University of California, Los Angeles; Cathy Stinear, PhD, Principal Investigator — University of Auckland, New Zealand; Achala Vagal, MD, Principal Investigator — University of Cincinnati
Locations (45):
- United States (45):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Banner University Medical Center, Tucson, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Kaiser Permanente Redwood City Medical Center, Redwood City, California
  - San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Heath Butterworth Hospital, Grand Rapids, Michigan
  - Mayo Clinic Saint Marys Campus, Rochester, Minnesota
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - The Mount Sinai Hospital, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Hospital, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - UVA Medical Center, Charlottesville, Virginia
  - Richmond VA Medical Center, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Wisconsin University Hospital, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Information about the study. — https://theverifystudy.com/